CLINICAL TRIAL: NCT02369497
Title: Ascension® Humeral Resurfacing Arthroplasty HRA Follow-Up Study
Brief Title: Ascension® Humeral Resurfacing Arthroplasty (HRA) Follow-Up Study
Acronym: HRA
Status: Terminated | Type: Observational
Why Stopped: PI left institution and site did not have resources to continue study
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-HRA-001
Record Dates: First submitted 2014-11-04; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary cohort: Primary cohort of subjects who receive the HRA device.
  Interventions: Device: HRA

INTERVENTIONS:
Device: HRA — Humeral head resurfacing with the HRA device

SUMMARY:
This is a prospective study on the Ascension HRA device to collect data to assess the safety and effectiveness of the HRA.

DETAILED DESCRIPTION:
This study protocol will provide guidance to investigators wanting to perform a non-randomized, consecutive enrollment, 10-year follow-up study of patients who are treated with the Ascension® HRA. Its purpose is to measure and document the outcomes associated with implanting the Ascension HRA prosthesis. Patients will be periodically assessed to collect data related to safety and effectiveness endpoints at the following intervals: preoperative, surgery/immediate post-op, 3 months, 6 months, 1 year, 2 year, 5 year, and 10 years.

ELIGIBILITY:
Inclusion Criteria:

Any patient who is to be treated with the Ascension HRA is eligible for inclusion in this study. Therefore, Principal Investigators should attempt to recruit all patients at the study site who are treated with the Ascension HRA

The following patient will be included in the study - Patient who:

* Is treated with the Ascension HRA
* Is disabled by either non-inflammatory or inflammatory arthritis (i.e. rheumatoid arthritis, osteoarthritis and avascular necrosis
* Has mild or moderate humeral head deformity and /or limited motion
* Has post-traumatic arthritis
* Has an intact or reparable rotator cuff
* Has the means and ability to return for all required study visits
* Is willing to participate in the study
* Has signed an Informed Consent Form
* Is at least 18 years of age and skeletally mature at the time of surgery
* Is less than 75 years of age at the time of surgery

Exclusion Criteria:

* Infection, sepsis, and osteomyelitis
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Rapid joint destruction, marked bone loss or bone resorption apparent on X-ray
* Revision procedures where other devices or treatments have failed
* Refuses to be in the study; or does not have the means and ability to return for all required study visits
* Currently participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with arthritis requiring humeral resurfacing arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2007-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score | 2 years
  The American Shoulder and Elbow Score is a functional outcome tool that has been validated for various shoulder conditions

SECONDARY OUTCOMES:
Range of Motion | 2 years
  Assessment of range of motion in the shoulder
Visual Analog Scale for pain | 2 years
  Patient assessed score of pain in the shoulder
X-rays | 2 years
  X-rays are conducted to assess the location and placement of the HRA device in the shoulder
Adverse events | Surgery; 3 month, 6 month, 1 year and 2 years post-op
  assessment of any adverse events that occur during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Candi Langmaid, MPH, CCRP, Study Director — Integra LifeSciences
Locations (1):
- Bay Pines VA Healthcare System, Bay Pines, Florida, United States